CLINICAL TRIAL: NCT00405041
Title: A Two-Center, Phase II/III, Randomized, Double-Blind, Placebo-Controlled, Study, to Assess the Therapeutic Efficacy of a Dietary Ingredient in Patients With Herniated Lumbar Disc Causing Nerve Root Compression
Brief Title: Randomized Controlled Study to Assess the Efficacy of a Dietary Ingredient in Patients With Herniated Lumbar Disc Compression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Ory Keynan, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-06-OK-06-203-CTIL; 107/06
Record Dates: First submitted 2006-11-21; First posted 2006-11-29 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Herniated Disc
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (1):
- A (Experimental)
  Interventions: Dietary Supplement: Dietary supplement GVG 2

INTERVENTIONS:
Dietary Supplement: Dietary supplement GVG 2 — 2.670 g/day for 14 days
  Other Names: GAVMATINE(TM)

SUMMARY:
The objective of the study is to evaluate the efficacy of a neuroprotective dietary supplement in patients suffering from herniated lumbar disc causing nerve root compression.

DETAILED DESCRIPTION:
Herniated lumbar discs exert pressure on nerves in the spine leading to pain, numbness, tingling and weakness of the leg, sometimes termed "sciatica". This syndrome affects about 1-2% of the population, usually at the age of 30 to 50 (the prime working years) leading to significant economic impact.

Injuries of nerves can lead to degeneration of the parent nerve cells, the neurons. Recent evidence indicates that herniated lumbar disc exerts mechanical pressure on spinal nerve roots that leads to local ischemia and inflammation resulting in nerve injury (i.e. neurotrauma). This neurotrauma can lead to degeneration of the corresponding nerve cells (dorsal root ganglia sensory neurons and spinal cord motoneurons), resulting in persistent deficits in motor functions, sensation and pain. Enhancing nerve cell survival capabilities (i.e., neuroprotection), therefore, should prove a novel therapeutic strategy for slowing or preventing degeneration of neurons resulting from herniated lumbar disc compression. Yet, in spite of an intensive search, clinically effective and safe neuroprotective therapeutic is not available.

The active ingredient in the dietary/medical food supplement under study was discovered to be an efficacious neuroprotective agent. The original findings, confirmed by laboratories throughout the world, indicate that the active compound is unique as it acts at multiple molecular targets to exert its robust neuropeotective effects.

The active ingredient is found in many plant, fish and meet foodstuffs and is being used and sold as a food supplement and nutraceutical. Its use as a neuroprotective agent is patented and thus, it constitutes an ideal candidate for neuroprotective treatment in herniated lumbar disc and other spine skeletal pathologies causing nerve compression.

The safety of the dietary supplement under study was clearly demonstrated in a recent clinical trial. Results of the trial demonstrated improvement in the general health status and indicated efficacy in alleviating symptoms in participants with herniated lumbar disc and other spine skeletal pathologies causing nerve root compression.

The present study is randomized, double-blind, placebo-controlled trial designed to ascertain the therapeutic efficacy of the dietary supplement in participants with herniated lumbar disc causing nerve damage symptoms. The study is being conducted in two medical centers in Israel. Eighty participants are presently being recruited and are screened under strict inclusion and exclusion criteria. Eligible individuals are invited to participate after signing a detailed informed consent prior to beginning of the study. The participants are being assigned randomly to receive either the dietary ingredient or placebo in a blind fashion whereby neither the treating physician nor the participant are aware of the type of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with diagnosis of herniated lumbar disc with nerve root compression, up to 3 months from beginning of symptoms.
* Participants' age: 18 - 75 years.
* Participants diagnosed by: i) computerized tomography CT or magnetic resonance imaging (MRI) when necessary; ii) neurological sensorimotor functional examination; iii) standard motor power scale; iv) pain sensation scales including the multidimensional tools: the Visual Analogue Scale of Pain Intensity for back and leg pain, the McGill Pain Questionnaire, and the Oswestry Disability Index; and v) Quality of life assessment based on the SF-36 questionnaire.
* Women must be non-pregnant, non-lactating, or sterilized, or postmenopausal.
* Participants must give a signed informed consent.

Exclusion Criteria:

* Participants with any significant clinical, medical or surgical condition, such as: cardiovascular (including those with hypertension and treated with antihypertensive agents), pulmonary, hepatic, renal, immune, endocrine, metabolic, digestive, malignancy, or allergic.
* Participants with low back pain emanating from causes other than herniated lumbar disc.
* Participants with any neuromuscular diseases.
* Participants with any musculoskeletal diseases.
* Participants with any neurological diseases.
* Participants with any history of alcohol or substance abuse within the last 2 years.
* Participants with gastric ulcer history.
* Participants who took any experimental drug within 90 days prior to screening.
* Women who are pregnant or breast feeding.
* Participants participating in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Measurements of herniated lumbar disc-related symptoms including sensorimotor neurological functions and pain sensations. And measurements of general quality of life based on the SF-36 questionnaire. | Within 14 days of treatment and follow-up at 30 and 60 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Dekel, M.D., Study Director — Tel Aviv Souraski Medical Center; Ory Keynan, M.D., Principal Investigator — Tel Aviv Souraski Medical Center
Locations (1):
- Tel Aviv Souraski Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Keynan O, Mirovsky Y, Dekel S, Gilad VH, Gilad GM. Safety and Efficacy of Dietary Agmatine Sulfate in Lumbar Disc-associated Radiculopathy. An Open-label, Dose-escalating Study Followed by a Randomized, Double-blind, Placebo-controlled Trial. Pain Med. 2010 Mar;11(3):356-68. doi: 10.1111/j.1526-4637.2010.00808.x. PMID 20447305